CLINICAL TRIAL: NCT01616940
Title: Minority AIDS Initiative Retention and Re-Engagement Project: Peer Re-Engagement Project
Brief Title: Minority AIDS Initiative Retention and Re-Engagement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Care Resource (Unknown); The Brooklyn Hospital Center (Other); Puerto Rico Community Network for Clinical Research on AIDS (Other); Justice Resource Institute (Other); Kansas City Free Health Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: U69HA23262
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Peer support
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-of-care (No Intervention): Standard-of-care at 3 demonstration sites includes: HIV medical care, medical case management, and referral to substance abuse, mental health, and housing services.
- Enhanced Peer Intervention (Experimental): Provides emotional, informational, and instrumental peer support, in addition to Standard-of-Care.
  Interventions: Behavioral: Enhanced Peer Intervention

INTERVENTIONS:
Behavioral: Enhanced Peer Intervention — Eight 30-60 minute educational sessions with peer will occur in-person bi-weekly once participant is randomized to intervention:
  * Introduction and Assessment
  * HIV Transmission & Viral Life Cycle
  * Effective Communication and Self-Advocacy
  * Understanding Lab Values
  * HIV Medications
  * Drug Resistance & Adherence, and Understanding & Managing Side Effects
  * Disclosure and Stigma
  * Harm & Risk Reduction
  Weekly check-ins will be by phone or in-person over 12 months. Check-in questions/tasks:
  * Are any services needed?
  * Have referrals or appointments been made?
  * Does patient need accompaniment to a visit?
  * Connect patient with services as needed.
  * Appointment reminders.
  * Overall well-being?
  * Schedule next peer contact.
  Other Names: Peer Re-Engagement Project (PREP)
  Arms: Enhanced Peer Intervention

SUMMARY:
The purpose of this study is to determine whether an enhanced peer intervention is effective in retaining and re-engaging at-risk people of color living with HIV/AIDS into care.

DETAILED DESCRIPTION:
This is a multi-site longitudinal study of an enhanced peer intervention to re-engage and retain high-risk people of color living with HIV into HIV primary care and other needed medical or social services. Three demonstration sites are implementing programs in which peers are employed as part of the health care team. Peers are trained to conduct educational sessions, provide emotional support, help prepare for and accompany patients to appointments, and debrief after visits.

Study participants will be current or newly enrolled patients of three clinics: CARE Resources, in Miami FL, the PATH Program at Brooklyn Hospital in Brooklyn, NY, and PR CONCRA located in San Juan Puerto Rico who (1) have been out of care for 4 months or more or (2) present a need for substance abuse, mental health, or housing services.

Data will be collected at baseline and follow up (at six and twelve months) through client questionnaires, selected medical chart data (visit dates, laboratory tests and values) and intervention encounter forms on approximately 375 HIV positive adults. The data collected for this study will allow us to assess changes in: (a) retention in HIV primary care, (b) viral load suppression, (c) health-related quality of life, (d) self-efficacy, and (e) HIV knowledge that may be associated with an enhanced peer intervention.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive; AND
* Age 18 years or older; AND
* Identifies as belonging to one or more of the following racial/ethnic groups: American Indian or Alaskan Native, Asian, Black or African-American, Hispanic or Latino, native Hawaiian or other Pacific Islander; AND
* New patient to clinic (including newly-diagnosed) whose initial assessment or intake form indicates a need for substance abuse treatment, mental health or housing services, or a past history of substance abuse or mental health services; OR
* The individual has been out of medical care at your clinic for 4 months or more.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of participants retained continuously in quality HIV care | 1 year
  "In HIV care" is defined as having a medical visit with a provider with prescribing privileges in an HIV care setting two or more times at least 3 months apart during the measurement year (HAB Performance Measure and National AIDS Strategy).
Number of participants who are virally suppressed | 1 year

SECONDARY OUTCOMES:
Change from Baseline in Health-related Quality of Life | 1 year
  Health-related quality of life will be measured using the SF-8 Health Survey by QualityMetric Incorporated.
Change from Baseline in Self-Efficacy | 1 year
  This will be measured using a scale that was developed and tested for the Chronic Disease Self-Management study*.
  * Lorig, K., Stewart, A., Ritter, P., Gonzalez, V., Laurent, D. & Lynch, J. (1996). Outcome Measures for Health Education and other Health Care Interventions. Thousand Oaks CA: Sage Publications, 24-25, 41-45.
Change from Baseline in HIV knowledge | 1 year
  HIV Knowledge will be measured using The HIV Treatment Knowledge Scale*.
  *Balfour, L., MacPherson, P., Garber, G., Beique, L. & Cameron, D. (2007). Development and psychometric validation of the HIV Treatment Knowledge Scale. AIDS Care, 19, 1141-1148.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Fox, MPH, Principal Investigator — Center for Advancing Health Policy and Practice, Boston University School of Public Health; Serena Rajabiun, MA, MPH, Principal Investigator — Center for Advancing Health Policy and Practice, Boston University School of Public Health; Howard Cabral, MPH, PhD, Principal Investigator — Department of Biostatistics, Boston University School of Public Health
Locations (4):
- United States (3):
  - Care Resource, Miami, Florida
  - Center for Advancing Health Policy and Practice, Boston, Massachusetts
  - PATH Center, The Brooklyn Hospital, Brooklyn, New York
- Puerto Rico Community Network for Clinical Research on AIDS, San Juan, Puerto Rico

REFERENCES:
- [Derived] Cabral HJ, Davis-Plourde K, Sarango M, Fox J, Palmisano J, Rajabiun S. Peer Support and the HIV Continuum of Care: Results from a Multi-Site Randomized Clinical Trial in Three Urban Clinics in the United States. AIDS Behav. 2018 Aug;22(8):2627-2639. doi: 10.1007/s10461-017-1999-8. PMID 29306990